CLINICAL TRIAL: NCT07381049
Title: Effect of Cash Benefits on Health Care Spending
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Brigham and Women's Hospital (Other); University of Michigan (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Sumit Agarwal, Primary Care Physician, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021P003354
Record Dates: First submitted 2026-01-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Health Care Costs; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in the treatment group received up to $400 per month.
  Interventions: Other: Cash Benefit
- Control Group (Active Comparator): Participants in the control group did not receive monthly cash benefits.
  Interventions: Other: No Cash Benefit

INTERVENTIONS:
Other: Cash Benefit — Spending from the cards was not restricted to food but could be spent on anything and anywhere Visa was accepted. The debit cards were credited with the first payment on November 18th, 2020 and the second payment on December 18th, 2020. The program continued with monthly credits through August 2021.
  Other Names: Cash Transfer; Debit Card; Guaranteed Income
  Arms: Treatment Group
Other: No Cash Benefit — No monthly cash benefit.
  Arms: Control Group

SUMMARY:
During the first two years of the COVID-19 pandemic, the City of Chelsea, Massachusetts held a lottery to allocate monthly cash benefits to its residents. Using data from the Chelsea Eats program, the investigators propose to study the impact of the cash benefit on health care spending.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Chelsea, Massachusetts
* Household income at or below 30% of the U.S. Department of Housing and Urban Development's Area Median Income

Exclusion Criteria:

* See inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3615 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Health care spending for medical services | 9 months
  Total payments to providers for medical services

SECONDARY OUTCOMES:
Health care spending in acute care setting | 9 months
  Total payments to providers for medical services in the acute care setting
Health care spending in outpatient setting | 9 months
  Total payments to providers for medical services in outpatient setting
Health care spending for prescription drugs | 9 months
  Total payments for prescription services

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Brigham and Women's Hospital / Harvard Medical School, Boston, Massachusetts
  - Harvard University, Cambridge, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT07381049/Prot_SAP_000.pdf